CLINICAL TRIAL: NCT03084575
Title: The Role of Selective Thermal Radiofrequency Saddle Rhizotomy In Managing Interactable Malignant Perineal Pain: A Comparative Study
Brief Title: Thermal Radiofrequency Versus Neurolytic Saddle Rhizotomyfor Severe Pereneal Cancer Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dina Nabil Abbas, Assistant professor of anethesia and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB No.201516026.2
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Interactable Malignant Perineal Pain
Keywords: neuroaxial rhizolysis -selective rhizolysis-thermal radiofrequency
MeSH Terms: interventions — Glycerol

STUDY DESIGN:
Intervention Model Description: randomization was done using a computer-generated random numbers with proper concealment in opaque sealed envelopes .
Who Masked: Outcomes Assessor
Masking Description: assessment will be done by junior stuff who is blind to the technique of intervention
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thermal Radiofrequency group (Active Comparator): Group 1 "RF group": in which patients will receive thermal radio Frequency, selective (unilateral S3, bilateral S4 and S5) saddle rhizotomy.
  Interventions: Procedure: Thermal radio Frequency, selective (unilateral S3, bilateral S4 and S5) saddle rhizotomy; Device: Thermal RF lesioning is done using Bailys RF generator
- phenol group (Active Comparator): Group 2 "phenol group": in which patients will recieve hyperbaric chemical saddle rhizotomy using 6% phenol in glycerin.
  Interventions: Drug: hyperbaric chemical saddle Rhizotomy (6 % pherol in glycerin)

INTERVENTIONS:
Procedure: Thermal radio Frequency, selective (unilateral S3, bilateral S4 and S5) saddle rhizotomy — Thermal RF lesioning is done using Bailys RF generator. TRF parameters are 80 C, 120 seconds the TRF lesion is repeated after 180 rotation of the needle tip again after sensory and motor pre-stimulation.
  Arms: Thermal Radiofrequency group
Drug: hyperbaric chemical saddle Rhizotomy (6 % pherol in glycerin) — L5-S1 intrathecal injection of 0.5-1 ml of 6 % pherol in glycerin. The patient is seated in the sitting position with 30-45o leaning backwards to make the posterior sensory roots lowermost.
  Other Names: 6 % pherol in glycerin
  Arms: phenol group
Device: Thermal RF lesioning is done using Bailys RF generator
  Arms: Thermal Radiofrequency group

SUMMARY:
The control of perineal malignant pain is difficult and challenging for pain physicians. Different modalities have been tried to treat this complex pain syndrome including pharmacotherapy and interventional therapy.

Neuroaxial phenol rhizolysis is simple and cheap option. However; for patients with pelvic or rectal neoplasms and intact bowel and bladder sphincteric functions, there are neurosurgical recomendations of selective sacral nerve roots rhizotomy blockade "as an alternative to chemical saddle rhizotomy".

DETAILED DESCRIPTION:
40 selected patients were randomly allocated into 2 groups "20 patients each"

Group 1 "RF group": in which patients underwent thermal radio Frequency, selective (unilateral S3, bilateral S4 and S5) saddle rhizotomy.

Group 2 "phenol group": in which patients underwent hyperbaric chemical saddle rhizotomy using 6% phenol in glycerin.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with moderate to severe perineal pain (VAS > 40mm over 100 mm scale).
* Intractable pain not responding to adequate tolerated opioid therapy + adjuvant therapy after reasonable period of time for at least 4 weeks (Rad and Kallmes, 2011).
* Limited life expectancy < 12 months (Slatakin etal 2003).
* Patients are continent to urine and stool (no stomas).

Exclusion Criteria:

* Uncorrected coagulopathy.
* Local or systemic sepsis.
* Known allergy to the used medications.
* Distorted local anatomy e.g. by advanced local neoplastic growth rendering the procedure technically difficult or hazardous.
* Sign of increased intracranial tension (Mintzer and Devarajan, 2012).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in VAS | baseline, one month, 3months
  VAS: A 100mm scale, horizontal line with 2 stop ends; the left end means no pain & the right end means the worst impaginable pain. It is a valid and practical scale for assessing chronic pain and for pain researches.
Functional improvement | baseline, one month, 3 months
  Functional improvement. It is a self-reported analysis for the primary outcome after performing pain interventions. It is divided into four categorie (0-25%) ≈ no or minimal functional improvement, (> 25% to 50%) ≈ mild improvement, (>50% to 75%) ≈ moderate improvement, and (>75% to 100%) ≈ marked improvement
Change in dose of daily drug consuption | base line, one month, 3 months
  drug (opioid, pregabalin & amitryptiline) consumption (mg/day) .

SECONDARY OUTCOMES:
ODI | baseline, one month, 3 months
  (Oswestry Disability Index): Self-reported questionnaire with 10 sections each with five items designed to assess limitations of various asctivities of daily living.
PGIC | baseline, one month and 3 months
  Patient satisfaction (PGIC): Patient Global Impression of Changes

CONTACTS AND LOCATIONS:
Overall Officials: Dina N Abbas, MD, Principal Investigator — National Cancer Institute,Cairo University

IPD SHARING:
Plan to Share IPD: Undecided